CLINICAL TRIAL: NCT04890743
Title: Effectiveness of Various Electrotherapy Methods in Treating People With Cervical Spine Pain Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Jolanta Zwolińska, PhD, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Urzeszow Club of Physical
Record Dates: First submitted 2021-04-29; First posted 2021-05-18 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2021-10

CONDITIONS: Cervical Spine Syndrome
Keywords: Cervical spine; Pain syndrome; Electrotherapy; TENS; Träbert ultrastimulation
MeSH Terms: conditions — Somatoform Disorders | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: The study will include healthy volunteers, students of the university in the area of Rzeszów with cervical spine pain syndrome caused by distance learning.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants of all 4 groups will benefit from a unified kinesiotherapeutic program. Then, after the randomization, participants will undergo treatments, but they will not know what type of therapy they will undergo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional TENS group (Experimental): One of the four groups created during randomization will undergo a unified program of kinesiotherapy and electrotherapy (Conventional TENS method).
  Interventions: Other: Kinesiotherapy combined with electrotherapy (Convenctional TENS method).
- Pseudo-acupuncture TENS group (Experimental): One of the four groups created during randomization will undergo a unified program of kinesiotherapy and electrotherapy (Pseudo-acupuncture TENS method).
  Interventions: Other: Kinesiotherapy combined with electrotherapy (Pseudo-acupuncture TENS method).
- Trabert ultrastimulation group (Experimental): One of the four groups created during randomization will undergo a unified program of kinesiotherapy and electrotherapy (Trabert ultrastimulation method).
  Interventions: Other: Kinesiotherapy combined with electrotherapy (Trabert ultrastimulation method)
- Placebo group (Placebo Comparator): One of the four groups created during randomization will undergo a unified program of kinesiotherapy and placebo electrotherapy.
  Interventions: Other: Kinesiotherapy combined with placebo electrotherapy

INTERVENTIONS:
Other: Kinesiotherapy combined with electrotherapy (Convenctional TENS method). — One of the four groups created during randomization will undergo a unified program of kinesiotherapy and electrotherapy (Conventional TENS method).
  Arms: Conventional TENS group
Other: Kinesiotherapy combined with electrotherapy (Pseudo-acupuncture TENS method). — One of the four groups created during randomization will undergo a unified program of kinesiotherapy and electrotherapy (Pseudo-acupuncture TENS method).
  Arms: Pseudo-acupuncture TENS group
Other: Kinesiotherapy combined with electrotherapy (Trabert ultrastimulation method) — One of the four groups created during randomization will undergo a unified program of kinesiotherapy and electrotherapy (Trabert ultrastimulation method).
  Arms: Trabert ultrastimulation group
Other: Kinesiotherapy combined with placebo electrotherapy — One of the four groups created during randomization will undergo a unified program of kinesiotherapy and placebo electrotherapy.
  Arms: Placebo group

SUMMARY:
Volunteers will take part in the study; Students of the university in the area of Rzeszow reporting chronic spinal ailments participation in remote learning. Applicant participants will be randomised into 3 groups of subjected to various electrotherapy procedures.

DETAILED DESCRIPTION:
Study participants will be tested:

1. Before a series of electrotherapy treatments.
2. 7 to 10 days after the end of electrotherapy.
3. 3 months after the end of electrotherapy. The study will use

   1. a self-authored survey taking into account: basic personal data (age, gender, value and BMI, lifestyle and degree of load on the cervical spine), information on the nature, intensity and frequency of the presence of pain in the spine cervical system, taking into account possible adverse reactions
   2. a questionnaire for subcjective assessment of the state of the spine Neck Disability Index,
   3. measuring the tone of the vertebral muscles in the cervical (myotonometer),
   4. a visual analog scale used to assess the severity of symptoms (Visual Analog Scale -VAS) Intervention;

   <!-- -->

   1. irradiation of the neck area with a sollux lamp with a blue filter
   2. individual exercises conducted according to the prepared author's mobility improvement program
   3. electrotherapy treatments:

      * Trabert currents
      * TENS currents (conventional)
      * TENS currents (pseudo-acupuncture)

ELIGIBILITY:
Inclusion Criteria:

* informed written consent of the patient to participate in the study
* no contraindications to electrotherapy in the area of the cervical spine;

Exclusion Criteria:

* poor tolerance of electrotherapy treatments;
* breaks between consecutive treatments longer than 3 days;
* failure to complete a series of kinesiotherapy and electrotherapy treatments;
* use of any stimulants during the observation period.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 1. Before a series of electrotherapy treatments.
  A questionnaire for subcjective assessment of the state of the spine.
Neck Disability Index | 2. 7 to 10 days after the end of electrotherapy.
  A questionnaire for subcjective assessment of the state of the spine.
Neck Disability Index | 3. 3 months after the end of electrotherapy.
  A questionnaire for subcjective assessment of the state of the spine.
Myotonometer | 1. Before a series of electrotherapy treatments.
  Measuring the tone of the vertebral muscles in the cervical.
Myotonometer | 2. 7 to 10 days after the end of electrotherapy.
  Measuring the tone of the vertebral muscles in the cervical.
Myotonometer | 3. 3 months after the end of electrotherapy.
  Measuring the tone of the vertebral muscles in the cervical.
Visual Analog Scale | 1. Before a series of electrotherapy treatments.
  A Visual Analog Scale used to assess the severity of symptoms. It enables the Patient to fine-tune the pain level on a scale from 0 to 10, where 0 is no pain at all and 10 is the maximum imaginable.
Visual Analog Scale | 2. 7 to 10 days after the end of electrotherapy.
  A Visual Analog Scale used to assess the severity of symptoms. It enables the Patient to fine-tune the pain level on a scale from 0 to 10, where 0 is no pain at all and 10 is the maximum imaginable.
Visual Analog Scale | 3. 3 months after the end of electrotherapy.
  A Visual Analog Scale used to assess the severity of symptoms. It enables the Patient to fine-tune the pain level on a scale from 0 to 10, where 0 is no pain at all and 10 is the maximum imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Perenc, docent prof, Study Director — University of Rzeszow
Locations (1):
- Laboratorium Czynników Fizykalnych w Rehabilitacji w Przyrodniczo-Medycznym Centrum Badań Innowacyjnych Uniwersytetu Rzeszowskiego, Rzeszów, Podkarpackie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Result] Martimbianco ALC, Porfirio GJ, Pacheco RL, Torloni MR, Riera R. Transcutaneous electrical nerve stimulation (TENS) for chronic neck pain. Cochrane Database Syst Rev. 2019 Dec 12;12(12):CD011927. doi: 10.1002/14651858.CD011927.pub2. PMID 31830313
- [Result] Martins-de-Sousa PH, Guimaraes Almeida MQ, da Silva Junior JM, Santos AS, Costa Araujo GG, de Oliveira Pires F, Fidelis-de-Paula-Gomes CA, Koga Ferreira VT, Dibai-Filho AV. Program of therapeutic exercises associated with electrotherapy in patients with chronic neck pain: Protocol for a randomized controlled trial. J Bodyw Mov Ther. 2020 Jan;24(1):25-30. doi: 10.1016/j.jbmt.2019.04.008. Epub 2019 Apr 25. PMID 31987553
- See also: Review of clinical trials assessing the effectiveness of exercise therapy and electrotherapy. — https://pubmed.ncbi.nlm.nih.gov/25659245/
- See also: In the study included adults with chronic neck pain (lasting > 12 weeks) that compared TENS alone or in combination with other treatments versus active or inactive treatments. The primary outcomes were pain, disability and adverse events. — https://pubmed.ncbi.nlm.nih.gov/31830313/
- See also: The objective of this study will be to evaluate the clinical effects of adding high- and low-frequency transcutaneous electrical nerve stimulation (TENS) in a program of specific therapeutic exercises for the treatment of patients with chronic neck pain. — https://pubmed.ncbi.nlm.nih.gov/31987553/